CLINICAL TRIAL: NCT02410707
Title: Adjunctive Nitrous Oxide During Emergency Department Propofol Sedation in Adults, a Pilot Study
Brief Title: Adjunctive Nitrous Oxide During Emergency Department Propofol Sedation in Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Albert Einstein Healthcare Network (Other)
Responsible Party: Principal Investigator, Joseph Herres, Principle Investigator, Albert Einstein Healthcare Network
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HN4641
Record Dates: First submitted 2015-02-11; First posted 2015-04-08 (Estimated); Results first posted 2020-04-08 (Actual); Last update posted 2020-04-08 (Actual); Status verified 2020-03

CONDITIONS: Joint Dislocation; Perianal Abscess; Abscess
Keywords: procedural sedation; procedural pain; procedural anxiolysis
MeSH Terms: conditions — Joint Dislocations; Abscess; Pain, Procedural | interventions — Nitrous Oxide; Propofol; Oxygen

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Nitrous Oxide Arm (Experimental): Patients undergoing procedural sedation with propofol will undergo an initial medical assessment including the history, physical examination, and vital signs. The patients will then receive Nitrous Oxide gas via a gas mixer device before receiving propofol. The device will mix and deliver nitrous oxide and oxygen in a 1:1 ratio, at a fixed concentration of 50%/50%. The on demand valve requires patient inspiration to trigger dosing.
  Interventions: Drug: Nitrous Oxide arm; Drug: Propofol; Drug: Oxygen

INTERVENTIONS:
Drug: Nitrous Oxide arm — Patients undergoing procedural sedation with propofol will undergo an initial medical assessment including the history, physical examination, and vital signs. The patients will then receive Nitrous Oxide gas via a gas mixer device before receiving propofol. The device will mix and deliver nitrous oxide and oxygen in a 1:1 ratio, at a fixed concentration of 50%/50%. The on demand valve requires patient inspiration to trigger dosing.
  Other Names: Nitrous Oxide; Sedera Gas Mixer; Propofol Sedation; Procedural Sedation
Drug: Propofol — The loading dose of propofol will be administered immediately after nitrous oxide discontinuation. All sedations in this trial will use propofol 1.0 mg/Kg initial dose, with 0.5 mg/Kg doses titrated to deep sedation. Once the patient is deeply sedated, the procedure will begin.
  Other Names: Diprivan
Drug: Oxygen — If pulse oximetry declines to less than 92%, subject will be placed on nasal cannula with administration of 2 liter flow of oxygen and titrated in increments of 1 L flow to maintain pulse oximetry greater than 92%
  Other Names: O2

SUMMARY:
The purpose of this study is to describe the safety and efficacy of nitrous oxide administration for pain and anxiety before propofol in patients requiring any procedure under sedation in the Emergency Department. Procedural sedation is the use of sedative, analgesic, and/or dissociative agents to relieve anxiety and pain associated with diagnostic and therapeutic procedures. Propofol is commonly used and is a sedative and amnestic, but provides no analgesia. Short acting opioids may be used for pain relief, but come with the risk of respiratory depression. An optimum analgesic to relieve pain in patients who need procedural sedation should be short acting, easy to administer and safe. Nitrous oxide may be a suitable agent, but literature supporting or rejecting its use in adults is lacking. This study aims to fill this gap. Adult patients capable of consenting, coming to the Emergency Department with painful condition requiring procedural sedation are the targeted population. Eligible patients who consent to the study will receive Nitrous Oxide gas delivered through a hand held mask before they receive propofol for the procedure. Information regarding their vitals, pain scores and medical condition will also be collected.

DETAILED DESCRIPTION:
This pilot study will be conducted in a prospective, non-randomized fashion using a convenience sample of 100 subjects undergoing sedation for Emergency Department procedures.

Recruitment Methods The research associates as well as the health care team (both residents and attending physicians) will screen patients who may need procedural sedation in the Emergency Department and may qualify for the study. Research associates will use the Medical Record

Procedures Involved in the Research Initial medical assessment will be made in accordance with established clinical procedures, including the history, physical examination, and vital signs. If by clinical assessment the patient meets eligibility criteria, then they will be approached by a research associate for enrollment in the study. After informed consent is obtained and prior to starting the sedation, standard vital sign monitoring will be placed on the patient (electrocardiogram, non-invasive blood pressure monitoring, pulse oximetry, and capnography). Level of consciousness will be determined using the modified Ramsay scale, which will be assessed at baseline. The Entitled Carbon Di Oxide (CO2) monitor will be used as the primary device to measure Entitled Carbon Di Oxide (CO2), with a nasal cannula capable of delivering supplemental oxygen and measuring Entitled CO2.

The Nitrous Oxide gas mixer system will be used as the primary nitrous oxide delivery device. It will mix and deliver nitrous oxide and oxygen in a 1:1 ratio, at a fixed concentration of 50%/50%. It uses a patient driven demand valve system that is hand held. This device provides a consistent, fixed 50%/50% blend of nitrous oxide (N2O) and oxygen (O2), eliminates the need to titrate, and provides fixed concentrations for controlled and consistent dosing. The device comparator detects dosing imbalance to protect against hypoxic mixtures, it cannot deliver nitrous gas without concurrent oxygen, and the device has an anti-asphyxia valve override. The on demand valve requires patient inspiration to trigger dosing. This portable device scavenges exhaled waste gases for environmental safety, as well as a key mechanism that renders the system inoperable without it for security.

After informed consent, the patient will fill out a pre procedure questionnaire and a 100 mm VAS baseline pain scale. The patient will be given the mask for delivery of nitrous oxide, and instructed on its use. The research associate will mark the time the patient began using the device electronically. Once IV access is established, and the team and patient are ready to begin the procedure, the nitrous oxide mask will be removed, and a 100% non rebreather mask delivering 15 liters a minute of supplemental oxygen will be placed on the patients face. The loading dose of propofol will then be administered immediately. All sedations in this trial will use propofol 1.0 mg/Kg initial dose, with 0.5 mg/Kg doses titrated to deep sedation. Once the patient is deeply sedated, the procedure will begin.

The subject's clinical data and sedation information (refer to data management) will be entered into a standardized data collection form. The data will be continuously recorded throughout the sedation and recovery periods. Study will end when the subjects recovers back to baseline mental status.

Vital signs will be flagged electronically when a physician intervenes for clinical respiratory depression. Respiratory depression will be defined as peripheral Oxygen saturation below 92%, Entitled CO2 level above 50, a rise or decrease of 10% above or below baseline, the loss of the Entitled CO2 waveform for more than 15 seconds. Level of consciousness will be determined using the modified Ramsay scale, which will be recorded at baseline and at the point of deepest sedation. Once the procedure is complete, and the patient is deemed back to their mental status baseline, they will fill out a post procedure satisfaction questionnaire, and a 100 mm VAS scale. They will be asked about procedure recall. The physician and nurse involved will also fill out a post procedure questionnaire.

System for screening, and they will be in charge of informed consent, enrollment, placement of the capnography monitor, as well as data collection. The health care team will be in charge of the procedural sedation and all other management.

ELIGIBILITY:
Inclusion Criteria:

* Spontaneous respirations
* 18 years of age and older
* American Society of Anesthesiologists (ASA) Physical Status Classification 1 or 2, who will be receiving sedation for an Emergency Department procedure.
* Ability to provide informed consent.

Exclusion Criteria:

* Comorbidities that affect ventilation, perfusion, or metabolism
* Intubated
* Cardiopulmonary instability
* Major trauma
* Sepsis
* American Society of Anesthesiologists (ASA) class 3, 4, and 5.
* Inability to provide informed consent
* Nursing home residents
* Age less than 18 years
* Non English speaking
* Pregnant women
* Under police custody

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2015-02; Primary Completion 2018-02 (Actual); Study Completion 2018-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Herres, DO, Principal Investigator — Albert Einstein Medical Center
Locations (1):
- Albert Einstein Medical Center, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Nitrous Oxide Arm: Patients undergoing procedural sedation with propofol will undergo an initial medical assessment including the history, physical examination, and vital signs. The patients will then receive Nitrous Oxide gas via a gas mixer device before receiving propofol. The device will mix and deliver nitrous oxide and oxygen in a 1:1 ratio, at a fixed concentration of 50%/50%. The on demand valve requires patient inspiration to trigger dosing.
  Nitrous Oxide arm: Patients undergoing procedural sedation with propofol will undergo an initial medical assessment including the history, physical examination, and vital signs. The patients will then receive Nitrous Oxide gas via a gas mixer device before receiving propofol. The device will mix and deliver nitrous oxide and oxygen in a 1:1 ratio, at a fixed concentration of 50%/50%. The on demand valve requires patient inspiration to trigger dosing.
  Propofol: The loading dose of propofol will be administered immediately after nitrous oxide use
Period: Overall Study
Arm/Group | Nitrous Oxide Arm
Started | 43
Completed | 43
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Nitrous Oxide Arm
Number analyzed (Participants) | 43
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.33 (20.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16
  Male | 27
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 10
  White | 22
  More than one race | 0
  Unknown or Not Reported | 11
Region of Enrollment [Number; unit: participants]
  United States | 43
Fracture/Reduction [Count of Participants; unit: Participants] | 41
Baseline VAS Pain Score [Mean (Standard Deviation); unit: units on a scale] — Visual Analog Scale (0-100mm), where 0 mm is minimum pain, and 100 mm is maximum pain.
  units on a scale | 76.29 (26.33)

OUTCOME MEASURES:

1. Primary Outcome: Total Number of Respiratory Depression Events
Description: End tidal CO2 and SpO2 measured every 20 milliseconds seconds captured by a monitoring device. Events of respiratory depression are defined as peripheral SaO2 below 92%, ETCO2 level above 50, a rise or decrease of 10% above or below baseline, and/or the loss of the ETCO2 waveform for more than 15 seconds
Time Frame: day 1
Measure: Number; unit: events
Arm/Group | Nitrous Oxide Arm
Number analyzed (Participants) | 43
events | 0

2. Secondary Outcome: Total Number of Airway Repositioning Events
Description: Presence or absence of physician intervention requiring airway repositioning by provider due to decreased oxygen saturation less than 92%
Time Frame: day 1
Measure: Number; unit: events of airway repositioning
Arm/Group | Nitrous Oxide Arm
Number analyzed (Participants) | 43
events of airway repositioning | 0

3. Secondary Outcome: Total Number of Events Requiring Additional Oxygen
Description: Presence or absence of physician intervention requiring additional oxygen via nasal cannula or non rebreather by the provider due to oxygen saturation less than 92%
Time Frame: day 1
Measure: Number; unit: events of additional oxygen
Arm/Group | Nitrous Oxide Arm
Number analyzed (Participants) | 43
events of additional oxygen | 0

4. Secondary Outcome: Total Number of Positive Pressure Ventilation Events
Description: Presence or absence of physician intervention requiring positive pressure ventilation via a bag valve max due to decreased oxygen saturation less than 92%
Time Frame: day 1
Measure: Number; unit: events of Positive pressure ventilation
Arm/Group | Nitrous Oxide Arm
Number analyzed (Participants) | 43
events of Positive pressure ventilation | 0

5. Secondary Outcome: Total Number of Endotracheal Intubation Events
Description: Presence or absence of physician intervention requiring endotracheal intubation by provider due to decreased oxygen saturation less than 92%
Time Frame: day 1
Measure: Number; unit: events of endotracheal intubation
Arm/Group | Nitrous Oxide Arm
Number analyzed (Participants) | 43
events of endotracheal intubation | 0

6. Secondary Outcome: Total Number of Physical Stimulation Events
Description: Presence or absence of physician intervention requiring physical stimulation by the provider due to decreased oxygen saturation less than 92%
Time Frame: day 1
Measure: Number; unit: number of subjects
Arm/Group | Nitrous Oxide Arm
Number analyzed (Participants) | 43
number of subjects | 2

7. Secondary Outcome: Patient, Physician, and Nurse Satisfaction Surveys
Description: Patient satisfaction with use of Nitrous Oxide in anxiolysis and pain control
Time Frame: day 1
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Arm/Group | Nitrous Oxide Arm
Number analyzed (Participants) | 43
percentage of subjects
  The number of subjects satisfied with the level of | 90 [71 to 97]
  The number of subjects would use NO in the future | 95 [77 to 99]
  Providers satisfied with the analgesia of NO | 82 [73 to 89]
  Providers ease of using NO device | 95 [77 to 99]
  Physicians would recommend use of NO | 95 [77 to 99]
  Nurses would recommend using NO device | 86 [65 to 95]
  Nurses felt it improved care | 76 [55 to 89]

8. Secondary Outcome: Post-Procedure VAS Pain Score
Description: Visual Analog Scale (0-100mm), where 0 mm is minimum pain, and 100 mm is maximum pain.
Time Frame: day 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Nitrous Oxide Arm
Number analyzed (Participants) | 43
units on a scale | 37.33 (32.63)

ADVERSE EVENTS:
Time Frame: 24 months
Description: Adverse events were defined by death, respiratory depression (hypoxia or increase in ETCO2), requiring airway intervention (oxygen, positive pressure ventilation, or endotracheal intubation).
Arm/Group | Nitrous Oxide Arm
All-Cause Mortality (participants affected / at risk) | 0/43
Serious Adverse Events (participants affected / at risk) | 0/43
Other Adverse Events (participants affected / at risk) | 0/43

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2014-07-01): https://cdn.clinicaltrials.gov/large-docs/07/NCT02410707/Prot_SAP_000.pdf